CLINICAL TRIAL: NCT02398279
Title: L-Arginine add-on Treatment for Schizophrenia: A Randomized, Double Blind, Placebo Controlled, Cross Over Study
Brief Title: L-arginine add-on Therapy in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, M. Kazim Yazici, Professor of Psychiatry, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 011D01101013
Record Dates: First submitted 2015-03-06; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; L-Arginine; nitric oxide; drug augmentation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Arginine-First (Experimental): For the first three weeks, L-Arginine 3 g bid (500mg capsules 6 x 2), one week wash-out, then for the next three weeks placebo capsules (6 x 2)
  Interventions: Dietary Supplement: L-Arginine; Other: Placebo
- Placebo-First (Experimental): For the first three weeks, placebo capsules (6 x 2), one week wash-out, then for the next three weeks L-Arginine 3 g bid (500 mg capsules 6 x 2)
  Interventions: Dietary Supplement: L-Arginine; Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-Arginine — Experimental supplement
Other: Placebo — Placebo capsules in the same color and shape with the experimental supplement

SUMMARY:
This study evaluates the addition of L-Arginine to the usual regimen in the treatment of schizophrenia in adults. As a requisite of crossover design, half of the participants started with L-Arginine and the other half with placebo and switched over after a three weeks use and one week of a washout period.

DETAILED DESCRIPTION:
L-arginine is the precursor of nitric oxide (NO), a neuromodulator of dopamine, gamma-aminobutyrate (GABA) and glutamate systems. Nitric oxide donors which increase NO levels at the cellular level could improve N-methyl-D-aspartate (NMDA) receptor dysfunction. Using L-arginine could bypass the blocked NMDA receptors and improve the therapeutic efficacy by reversing the dysfunction.

The investigators proposed that using L-Arginine, a dietary supplement in most cultures, might constitute a safe option as an add-on treatment which may display beneficial effects on positive, negative, cognitive and affective symptoms associated with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia-Schizoaffective Disorder
* Clinical Global Impression >4
* Able to take oral medication and likely to comply the required evaluations
* On stable medication regimen for 8 weeks
* Competent and willing to give informed consent

Exclusion Criteria:

* Uncontrolled medical illness (renal disease, hepatic, cardiac diseases, gout, asthma, diabetes, sickle cell anemia, low-high blood pressure)
* History of Myocardial Infarction (MI)
* History of genital herpes infections/ receiving lysine containing treatments
* Pregnancy/ lactation
* Substance related and Addictive Disorders
* Drugs that might induce hypotension
* Intolerance to L-arginine and ingredients of placebo or L-arginine capsule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale | baseline and week 3
  Evaluating change in Positive and Negative Syndrome Scale between baseline and Week 3, comparing subjects treated with L-Arginine for 3 weeks to subjects treated with placebo for 3 weeks.

SECONDARY OUTCOMES:
Change from baseline in Neuropsychological Test Battery | baseline and week 3
  Evaluating change in Neuropsychological Test Battery between baseline and Week 3, comparing subjects treated with L-Arginine for 3 weeks to subjects treated with placebo for 3 weeks.
Change from baseline in the The Calgary Depression Scale for Schizophrenia | baseline and week 3
  Evaluating change in The Calgary Depression Scale for Schizophrenia between baseline and Week 3, comparing subjects treated with L-Arginine for 3 weeks to subjects treated with placebo for 3 weeks.
Change from baseline in Clinical Global Impression - Severity | baseline and week 3
  Evaluating change in Clinical Global Impression - Severity between baseline and Week 3, comparing subjects treated with L-Arginine for 3 weeks to subjects treated with placebo for 3 weeks.
Change from baseline in Abnormal Involuntary Movement Scale | baseline and week 3
  Evaluating change in Abnormal Involuntary Movement Scale between baseline and Week 3, comparing subjects treated with L-Arginine for 3 weeks to subjects treated with placebo for 3 weeks.
Change from baseline in Uku Side Effects Rating Scale | baseline and week 3
  Evaluating change in Uku Side Effects Rating Scale between baseline and Week 3, comparing subjects treated with L-Arginine for 3 weeks to subjects treated with placebo for 3 weeks.
Change from baseline in blood pressure | baseline and week 7
Change from baseline in heart rate | baseline and week 7
Change from baseline in temperature | baseline and week 7
Change from baseline in respiratory rate | baseline and week 7
Change from baseline in weight | baseline and week 7
Change from baseline in electrocardiogram | baseline and week 7
Change from baseline in complete blood count | baseline and week 7
  Composed of different measures. Change in any measure indicates impairment in the composite measure
Change from baseline in alanine aminotransferase | baseline and week 7
Change from baseline in aspartate aminotransferase | baseline and week 7
Change from baseline in alkaline phosphatase | baseline and week 7
Change from baseline in urea | baseline and week 7
Change from baseline in creatinine | baseline and week 7
Change from baseline in sodium | baseline and week 7
Change from baseline in potassium | baseline and week 7
Change from baseline in chloride | baseline and week 7
Change from baseline in calcium | baseline and week 7
Change from baseline in thyroid-stimulating hormone | baseline and week 7
Change from baseline in free T4 | baseline and week 7
Change from baseline in total cholesterol | baseline and week 7
Change from baseline in HDL | baseline and week 7
Change from baseline in LDL | baseline and week 7
Change from baseline in triglycerides | baseline and week 7
Change from baseline in human chorionic gonadotropin | baseline and week 7
  Pregnancy test in women

CONTACTS AND LOCATIONS:
Overall Officials: Kazım M Yazıcı, MD, Principal Investigator — Hacettepe University Faculty of Medicine Department of Psychiatry
Locations (1):
- Hacettepe University Faculty of Medicine Department of Psychiatry, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Boger RH. The pharmacodynamics of L-arginine. J Nutr. 2007 Jun;137(6 Suppl 2):1650S-1655S. doi: 10.1093/jn/137.6.1650S. PMID 17513442
- [Background] Maia-de-Oliveira JP, Trzesniak C, Oliveira IR, Kempton MJ, Rezende TM, Iego S, Baker GB, Dursun SM, Machado-de-Sousa JP, Hallak JE. Nitric oxide plasma/serum levels in patients with schizophrenia: a systematic review and meta-analysis. Braz J Psychiatry. 2012 Oct;34 Suppl 2:S149-55. doi: 10.1016/j.rbp.2012.07.001. English, Portuguese. PMID 23429845
- [Background] Vayisoglu S, Anil Yagcioglu AE, Yagcioglu S, Karahan S, Karci O, Gurel SC, Yazici MK. Lamotrigine augmentation in patients with schizophrenia who show partial response to clozapine treatment. Schizophr Res. 2013 Jan;143(1):207-14. doi: 10.1016/j.schres.2012.11.006. Epub 2012 Dec 2. PMID 23217729
- [Derived] Kocyigit Y, Yoca G, Karahan S, Ayhan Y, Yazici MK. [L-Arginine Add-On Treatment for Schizophrenia: A Randomized,Double-Blind, Placebo-Controlled, Crossover Study]. Turk Psikiyatri Derg. 2018 Fall;29(3):147-153. Turkish. PMID 30260460